CLINICAL TRIAL: NCT04144998
Title: Substudy on Central Sensitization and Outcome of Endometriosis Surgery of the PROMPT Study
Brief Title: Central Sensitization and Outcome of Endometriosis Surgery
Status: Completed | Type: Observational
Sponsor: Benno Rehberg-Klug (Other)
Responsible Party: Sponsor-Investigator, Benno Rehberg-Klug, Dr. Benno Rehberg-Klug, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: EndoPROMPT
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: central sensitization inventory (questionnaire) — T.G. Mayer, R. Neblett, H. Cohen, et al. The development and psychometric validation of the central sensitization inventory Pain Pract, 12 (2012), pp. 276-285

SUMMARY:
This study will evaluate whether the degree of central sensitization as measured by the questionnaire "central sensitization inventory CSI" is related to the outcome of surgical endometriosis treatment

ELIGIBILITY:
Inclusion Criteria:

* Primary surgery because of pelvic/abdominal pain under suspected diagnosis of and with the aim to confirm endometriosis
* Elective abdominal surgery in women with pelvic/abdominal pain and confirmed endometriosis

Exclusion Criteria:

* Patient is unable to give consent
* Cognitive impairment
* Patient outcomes questionnaire is not available in a language that the patient knows.
* Secondary surgery due to complications
* Endometriosis Surgery due to infertility

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for elective endometriosis surgery
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
endometriosis health profile EHP-30 pain subscale | 6 months
  Pain subscale of the questionnaire "endometriosis health profile" EHP-30, scale from 0-100, higher values indicate worse health status

SECONDARY OUTCOMES:
other subscales of the endometriosis health profile EHP-30 | 6 months
  control and powerlessness scale, emotional well-being scale, social support scale, self-image scale, all scales from 0-100, higher values indicate worse health status

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided